CLINICAL TRIAL: NCT05764889
Title: Study on the Protective Effect of a Flexible Sleeve Penis Protection Device on Penis After Circumcision
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Liu Zhuo (Other)
Responsible Party: Sponsor-Investigator, Liu Zhuo, Attending Doctor, Peking University Third Hospital
Organization: Peking University Third Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: M2022628
Record Dates: First submitted 2023-02-09; First posted 2023-03-13 (Actual); Last update posted 2023-03-31 (Actual); Status verified 2023-03

CONDITIONS: Circumcision, Male
Keywords: Circumcision; Postoperative complications; Protection devices
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Intervention Model Description: Patients in the experimental group were wrapped with this device postoperatively Patients in the control group were wrapped with traditional gauze postoperatively.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): Patients in the experimental group were wrapped with the Flexible Sleeve Penis Protection Device post-operatively.
  Interventions: Other: wrapped with the Flexible Sleeve Penis Protection Device
- Control group (Other): Patients in the control group were wrapped with traditional gauze after operation.
  Interventions: Other: wrapped with traditional gauze

INTERVENTIONS:
Other: wrapped with the Flexible Sleeve Penis Protection Device — Patients in the experimental group were wrapped with the Flexible Sleeve Penis Protection Device post-operatively.
  Patients in the control group were wrapped with traditional gauze post-operatively.
  Arms: Experimental group
Other: wrapped with traditional gauze — Patients in the experimental group were wrapped with the Flexible Sleeve Penis Protection Device post-operatively.
  Patients in the control group were wrapped with traditional gauze post-operatively.
  Arms: Control group

SUMMARY:
Circumcision is a common clinical procedure for both circumcision and phimosis, which are common disorders of the male reproductive system. For post-circumcision patients, a flexible sleeve penile protection device was invented as a modification of the traditional gauze bandage. This study investigated the protective effect of the device by recruiting post-circumcision patients to use the device and collecting indicators related to post-operative recovery and patients' experience of using the device.

DETAILED DESCRIPTION:
Circumcision is a common clinical procedure for both circumcision and phimosis, which are common disorders of the male reproductive system. Post-circumcision patients remain at risk of gauze detachment, wound pain and post-operative bleeding, leading to serious post-operative adverse effects, including complications such as dehiscence and infection. The investigators have invented a flexible sleeve penile protection device, which consists of two components, a flexible sleeve and a hood, the main function of the flexible sleeve is to stop bleeding with compression and immobilisation, and the main function of the hood is to provide protection to the head of the penis and prevent the wound from rubbing against clothing leading to pain.

The aim of this study was to investigate the protective effect of a flexible sleeve penile protection device on post-circumcision patients in terms of gauze loosening and dislodging, post-operative pain and post-operative bleeding. This study was a prospective randomized controlled trial of patients who underwent circumcision at Peking University Third Hospital from February 2023 to May 2023. Patients in the experimental group were wrapped with this device postoperatively, while patients in the control group were wrapped with traditional gauze postoperatively. Patients were followed up regularly after surgery, and indicators such as complications, pain and recovery time were collected to investigate the protective effect of this device.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosed redundant prepuce and circumcised at Peking University Third Hospital.
2. Male patients aged between 12 and 60 years (inclusive).
3. The person or guardian fully understands and signs the informed consent form.

Exclusion Criteria:

1. Acute urinary and genital infections, such as acute urethritis, acute prostatitis, acute epididymitis, etc., or trauma.
2. Abnormal blood clotting function.
3. Those who are allergic to the materials used in the manufacture of the product.
4. Patients who are mentally incapable or unable to understand the requirements for participation in the study and have difficulty in cooperating.
5. Subjects who, in the opinion of the investigator, are unable to comply with follow-up, compromising the scientific validity and integrity of the study.

Ages: 12 Years to 60 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-03-15 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-07-30 (Estimated)

PRIMARY OUTCOMES:
Post-operative complication | through study completion, an average of 12weeks
  Assessing the incidence of post-operative complications
Foreskin edema score | through study completion, an average of 12weeks
  Assessment of foreskin oedema which includes 0-6 points. A higher score means a more severe case of penile foreskin oedema
Healing time | through study completion, an average of 12weeks
  Time for sutures to come off completely and time for wound healing

SECONDARY OUTCOMES:
Wound pain assessment | through study completion, an average of 12weeks
  Using the Visual analogue scale ，which includes 0-10 points. A higher score means more pain
Comfort and convenience assessment | through study completion, an average of 12weeks
  Comfort and convenience assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Zhuo Liu, MD, Study Director — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mu J, Fan L, Liu D, Zhu D. A Comparative Study on the Efficacy of Four Types of Circumcision for Elderly Males with Redundant Prepuce. Urol J. 2020 May 16;17(3):301-305. doi: 10.22037/uj.v0i0.4973. PMID 31364098
- [Background] Abara EO. Prepuce health and childhood circumcision: Choices in Canada. Can Urol Assoc J. 2017 Jan-Feb;11(1-2Suppl1):S55-S62. doi: 10.5489/cuaj.4447. PMID 28265321
- [Background] Soltany S, Ardestanizadeh A. The study of the factors affecting the time of ring fall off in circumcision using Plastibell. J Family Med Prim Care. 2020 Jun 30;9(6):2736-2740. doi: 10.4103/jfmpc.jfmpc_1261_19. eCollection 2020 Jun. PMID 32984117
- [Background] van den Dungen IAL, Rynja SP, Bosch JLHR, de Jong TPVM, de Kort LMO. Comparison of preputioplasty and circumcision in distal hypospadias correction: long-term follow-up. J Pediatr Urol. 2019 Feb;15(1):47.e1-47.e9. doi: 10.1016/j.jpurol.2018.08.001. Epub 2018 Aug 20. PMID 30270101